CLINICAL TRIAL: NCT07130331
Title: Efficacy and Influencing Factors Analysis of Secukinumab in Patients With Axial Spondyloarthritis in a Real-World Setting
Brief Title: Efficacy and Influencing Factors of Secukinumab in Patients With Axial Spondyloarthritis
Status: Completed | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0544-02
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Axial Spondylarthritis (axSpA); Secukinumab
Keywords: Axial spondyloarthritis; ASAS40
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with axial spondyloarthritis: Patients with axial spondyloarthritis
  Interventions: Drug: Secikinumab

INTERVENTIONS:
Drug: Secikinumab — secukinumab 150 mg at weeks 0, 1, 2, 3, and 4, followed by 150 mg s.c. every 4 weeks

SUMMARY:
This study aimed to explore the efficacy and influencing factors of secukinumab in axSpA patients by conducting a real-world retrospective analysis.

DETAILED DESCRIPTION:
Interleukin-17 (IL-17) plays a key role in axSpA joint inflammation, cartilage injury and bone remodeling.The 2022 ASAS-EULAR recommendations recommended the use of IL-17 inhibitors as first-line therapy for patients who have had an inadequate response to conventional agents including non-steroidal anti-inflammatory drugs (NSAIDs) and disease-modifying antirheumatic drugs (DMARDs). Secukinumab, a fully human monoclonal IgG1/κ antibody targeting IL-17A, was approved in the US in 2016 for the treatment of AS and in 2020 for the treatment of nr-axSpA. Although several studies have shown that secukinumab significantly reduces pain symptoms and diseases activity in axSpA patients, a significant proportion of patients experience treatment failure during the maintenance phase. This study aimed to explore the efficacy and influencing factors of secukinumab in axSpA patients by conducting a retrospective analysis in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the 2011 Assessment of SpondyloArthritis international Society (ASAS) classification criteria for axial spondyloarthritis
2. Treated with secukinumab with regular follow up
3. Patients who visited the Rheumatology clinic from Jun 2020 to Jul 2024 retrieved by Hospital Information System

Exclusion Criteria:

1. allergic to secukinumab
2. concomitant with other rheumatic immune diseases
3. patients with malignancies or serious infections
4. patients with poor compliance and lost to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult axSpA patients treated with Secukinumab
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
The Percentage of Participants Who Achieved an Assessment of Spondylo Arthritis International Society (ASAS) 40 Response | At week 12 after administration.
  Assessment of Spondylo Arthritis International Society criteria (ASAS) consist of 6 domains (4 main and 2 additional assessment domains): 1. Patient's global assessment measured on a NRS; 2. Patient's assessment of back pain, measured on a NRS; 3. Function represented by Bath Ankylosing Spondylitis Functional Index (BASFI) average of 10 questions as measured by NRS; 4. Inflammation represented by mean duration and severity of morning stiffness, on the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) as measured by NRS; 5. Spinal mobility represented by the Bath Ankylosing Spondylitis Metrology Index (BASMI) lateral spinal flexion assessment; 6. C-reactive protein (acute phase reactant).
  ASAS40 response is defined as an improvement of ≥40% and ≥2 units on a scale of 10 in at least three of the four ASAS main domains and no worsening at all in the remaining domain. A higher score on the NRS signifies higher severity.

OTHER OUTCOMES:
Laboratory parameters | At week 12 after administration
  White blood cell count, hemoglobin count, platelet count; level of lactate dehydrogenase, alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, creatinine, uric acid, e-GFR, albumin, globulin, erythrocyte sedimentation rate, C-reactive protein

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rudwaleit M, van der Heijde D, Landewe R, Akkoc N, Brandt J, Chou CT, Dougados M, Huang F, Gu J, Kirazli Y, Van den Bosch F, Olivieri I, Roussou E, Scarpato S, Sorensen IJ, Valle-Onate R, Weber U, Wei J, Sieper J. The Assessment of SpondyloArthritis International Society classification criteria for peripheral spondyloarthritis and for spondyloarthritis in general. Ann Rheum Dis. 2011 Jan;70(1):25-31. doi: 10.1136/ard.2010.133645. Epub 2010 Nov 24. PMID 21109520
- [Background] Marzo-Ortega H, Sieper J, Kivitz A, Blanco R, Cohen M, Martin R, Readie A, Richards HB, Porter B; Measure 2 Study Group. Secukinumab and Sustained Improvement in Signs and Symptoms of Patients With Active Ankylosing Spondylitis Through Two Years: Results From a Phase III Study. Arthritis Care Res (Hoboken). 2017 Jul;69(7):1020-1029. doi: 10.1002/acr.23233. Epub 2017 Jun 7. PMID 28235249
- [Background] Danve A, Deodhar A. Treatment of axial spondyloarthritis: an update. Nat Rev Rheumatol. 2022 Apr;18(4):205-216. doi: 10.1038/s41584-022-00761-z. Epub 2022 Mar 10. PMID 35273385
- [Background] Ramiro S, Nikiphorou E, Sepriano A, Ortolan A, Webers C, Baraliakos X, Landewe RBM, Van den Bosch FE, Boteva B, Bremander A, Carron P, Ciurea A, van Gaalen FA, Geher P, Gensler L, Hermann J, de Hooge M, Husakova M, Kiltz U, Lopez-Medina C, Machado PM, Marzo-Ortega H, Molto A, Navarro-Compan V, Nissen MJ, Pimentel-Santos FM, Poddubnyy D, Proft F, Rudwaleit M, Telkman M, Zhao SS, Ziade N, van der Heijde D. ASAS-EULAR recommendations for the management of axial spondyloarthritis: 2022 update. Ann Rheum Dis. 2023 Jan;82(1):19-34. doi: 10.1136/ard-2022-223296. Epub 2022 Oct 21. PMID 36270658
- [Background] McGonagle DG, McInnes IB, Kirkham BW, Sherlock J, Moots R. The role of IL-17A in axial spondyloarthritis and psoriatic arthritis: recent advances and controversies. Ann Rheum Dis. 2019 Sep;78(9):1167-1178. doi: 10.1136/annrheumdis-2019-215356. Epub 2019 Jul 5. PMID 31278139
- [Background] Taams LS, Steel KJA, Srenathan U, Burns LA, Kirkham BW. IL-17 in the immunopathogenesis of spondyloarthritis. Nat Rev Rheumatol. 2018 Aug;14(8):453-466. doi: 10.1038/s41584-018-0044-2. PMID 30006601
- [Background] Chyuan IT, Chen JY. Role of Interleukin- (IL-) 17 in the Pathogenesis and Targeted Therapies in Spondyloarthropathies. Mediators Inflamm. 2018 Feb 12;2018:2403935. doi: 10.1155/2018/2403935. eCollection 2018. PMID 29670461
- [Background] Zhao J, Huang C, Huang H, Pan JK, Zeng LF, Luo MH, Liang GH, Yang WY, Liu J. Prevalence of ankylosing spondylitis in a Chinese population: a systematic review and meta-analysis. Rheumatol Int. 2020 Jun;40(6):859-872. doi: 10.1007/s00296-020-04537-0. Epub 2020 Mar 3. PMID 32125505
- [Background] Rudwaleit M, van der Heijde D, Landewe R, Listing J, Akkoc N, Brandt J, Braun J, Chou CT, Collantes-Estevez E, Dougados M, Huang F, Gu J, Khan MA, Kirazli Y, Maksymowych WP, Mielants H, Sorensen IJ, Ozgocmen S, Roussou E, Valle-Onate R, Weber U, Wei J, Sieper J. The development of Assessment of SpondyloArthritis international Society classification criteria for axial spondyloarthritis (part II): validation and final selection. Ann Rheum Dis. 2009 Jun;68(6):777-83. doi: 10.1136/ard.2009.108233. Epub 2009 Mar 17. PMID 19297344
- [Background] Simone D, Al Mossawi MH, Bowness P. Progress in our understanding of the pathogenesis of ankylosing spondylitis. Rheumatology (Oxford). 2018 Aug 1;57(suppl_6):vi4-vi9. doi: 10.1093/rheumatology/key001. PMID 30445483